CLINICAL TRIAL: NCT01825382
Title: Role of Mobile Technology to Improve Diabetes Care in Adults With Type 1 Diabetes: the REMOTE-T1D Study, a Pilot Study
Acronym: REMOTE-T1D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sanofi (Industry); Colorado Prevention Center (Other)
Responsible Party: Principal Investigator, Satish K. Garg, Professor of Medicine and Pediatrics, Editor in Chief DT&T, University of Colorado, Denver
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REMOTE-T1D
Record Dates: First submitted 2013-01-29; First posted 2013-04-05 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Accu-chek Meter (No Intervention): Patients receiving the Accu-chek nano meter for use during the study.
- iBGStar meter interventional Arm (Experimental): Subjects are given iBGstar meter along with iPhone to use as interventional meter.
  Interventions: Device: iBGStar meter

INTERVENTIONS:
Device: iBGStar meter — Subjects will receive iBGStar meter and iPhone to use as meter during the study.
  Arms: iBGStar meter interventional Arm

SUMMARY:
The goal of this prospective pilot study is to evaluate the use of remote technology (iBGStar in combination with Diabetes Manager App on iPhone) to patient related outcomes, and a hypoglycemia fear questionnaire. In the future, this study might lead to investigating the role of social media with mobile phones in Type 1 Diabetes (T1D) care. Moreover, the number of patients with T1D continues to increase, and such technology could conceivably help compensate for the shortages of endocrinologists providing care.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, 'open-label,' investigator initiated pilot study evaluating the role of mobile technology to improve diabetes care in adults with type 1 diabetes (REMOTE-T1D). We hypothesize that the use of mobile technology (iBGStar® technology [iPhone® plus the BGStar®]) will result in improvement in Patient Reported Outcomes (PRO), and Treatment Satisfactions with a possible reductions of glucose excursions, A1c, and severe hypoglycemia as compared to routine clinical care using traditional glucose meter SMBG-Accu-chek®. This study aims to demonstrate the efficacy of these technologies in a clinical setting with a hope to improve outcomes and health care cost savings.

The study will enroll 100 patients from the Barbara Davis Center Adult clinic over the age of 18 years who will be randomized in a 1:1 fashion to intervention group using mobile technology (iBG Star) vs. continued routine clinical care (control) using SMBG-Accu-chek meter. All subjects will be followed for study visits with similar frequency at baseline, 1-week, 1-month, 3-months, and 6-months and wear a continuous glucose monitor (CGM) using a DexCom SEVEN Plus® system in a blinded mode for 7 days at baseline (wk0), 1mo, 3mo, and 6mo.

Laboratory analysis for A1c will be performed at baseline, 1-month 3-months, and 6-months. Routine blood tests will be performed in all subjects at baseline, 3months, and 6-months. Blinded CGM data will be analyzed for mean blood glucose values, time spent in hyperglycemic (>240, >300mg/dl) and hypoglycemic (<50, <70, <80 mg/dl) ranges and various indices of glycemic variability.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that meet the following criteria will be considered for admission to the study:

  1. Signed informed consent before any study-related activities
  2. Male or female aged 18 years and older T1D duration >1 year
  3. A1c <10%
  4. Willingness to routinely practice at least 3-7 blood glucose measurements per day
  5. Ability and willingness to adhere to the protocol including scheduled study visits and blinded CGM wear intermittently) for 6 months. During the weeks of blinded CGM wear, subjects will not be able to use their own real-time CGMs (if they own it)
  6. Able to speak, read and write English

Exclusion Criteria:

* Subjects will be excluded from the study if any of the following apply:

  1. Pregnant or intention to become pregnant during the course of the study
  2. Severe unexplained hypoglycemia requiring emergency treatment in the previous 6 months
  3. Use of systemic or inhaled corticosteroids
  4. History of hemoglobinopathies
  5. Diagnosis of anemia
  6. History of pancreatitis
  7. Extensive skin changes/diseases that inhibit wearing a sensor on normal skin
  8. Known allergy to adhesives
  9. Current participation in another investigational study protocol. Must have completed a previous study at least 30 days prior to enrollment.
  10. Any other condition, as determined by the investigator, which could make the subject unsuitable for the trial, impairs the subject's suitability for the trial, or impairs the validity of the informed consent
  11. Subjects will not be allowed to use real-time CGM during the blinded CGM wear week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes as it relates to hypoglycemia fear and quality of life. | 6 months
  Primary outcome is patient related outcomes and changes based on the hypoglycemia fear questionnaire and changes in patient comfort in meter use.

SECONDARY OUTCOMES:
Improvement in glucose control and indices off glucose variability from SMBG and CGM data. | 6 months
  Improvement in parameters of glycemic variability as measured by glucose excursions from SMBG and CGM downloads and various indices (J-index, mean amplitude of glycemic excursion (MAGE), high blood glucose index (HBGI), low blood glucose index (LBGI), from, CGM downloads. Reduction in A1c of 0.3% from screening to 3-months and maintained at 6-months, and reduction of hypoglycemia (measured or self reported). Cost analysis will be done based upon primary and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Satish K Garg, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

REFERENCES:
- [Derived] Garg SK, Shah VN, Akturk HK, Beatson C, Snell-Bergeon JK. Role of Mobile Technology to Improve Diabetes Care in Adults with Type 1 Diabetes: The Remote-T1D Study iBGStar(R) in Type 1 Diabetes Management. Diabetes Ther. 2017 Aug;8(4):811-819. doi: 10.1007/s13300-017-0272-5. Epub 2017 May 29. PMID 28555339